CLINICAL TRIAL: NCT05751057
Title: The Role of Cardiovascular Magnetic Resonance in Patients With Non-ST- Elevation- Myocardial Infarction: the TITAN-MRI Study
Brief Title: The Role of Cardiovascular Magnetic Resonance in Patients With Non-ST- Elevation- Myocardial Infarction
Acronym: TITAN-MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardiocentro Ticino (Other)
Responsible Party: Principal Investigator, Anna Giulia Pavon, Consultant Cardiologist, Cardiovascular Imaging Laboratory, Cardiocentro Ticino
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 01-TITAN-MRI
Record Dates: First submitted 2023-01-12; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Non-ST Elevation Myocardial Infarction (NSTEMI)
Keywords: cardiovascular magnetic resonance; Myocardial Infaction; Invasive Coronary Angiography
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NSTEMI patients (Experimental): Patients will undergo CMR before ICA
  Interventions: Diagnostic Test: Cardiovascular Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Cardiovascular Magnetic Resonance — All NSTEMI patients will undergo to CMR before invasive coronary intervention.

SUMMARY:
The goal of this prospective study is to evaluate the role of cardiovascular magnetic resonance (CMR) in patients with suspected non-ST elevation myocardial infarction (NSTEMI). The main endpoint is the reclassification rate, defined as the number of patients in whom the information provided by pre-angiography CMR affects the revascularization strategy or the final diagnosis.

Participants will undergo to CMR before invasive coronary angiography (ICA).

DETAILED DESCRIPTION:
All patients with NSTEMI eligible for the study undergo CMR prior to ICA. To avoid any delay in patients' treatment all examination will be analyzed by local trained staff at each center. All patients will thereafter undergo ICA and the standard of care (SOC) decision-making on revascularization strategy and diagnosis will be declared by the treating physician, which will be blinded to the participation of the patients in the study and about CMR results. The treating physician will also declare patient's next management according to ICA results. After having declared the diagnosis, the treating physician will then be informed about the CMR findings. Therefore, according to CMR results the treating physician may eventually modify the initial diagnosis and management. Treatment plan modifications include difference in the identification of the culprit lesion, referring the patient to medical therapy instead of a revascularization procedure or viceversa, switching from a percutaneous to a surgical revascularization procedure or viceversa, or need for further cardiac or non-cardiac investigations. Initial diagnosis includes confirmed NSTEMI or all other possible alternative diagnosis and proposed additional diagnostic examination(s) for further differential diagnosis.

The CMR-modified SOC (CMR-SOC) and diagnosis made considering CMR results will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Presence of criteria for acute myocardial infarction according to the Fourth Universal Definition of Myocardial Infarction:
* Signs and symptoms of myocardial ischemia
* Detection of acute myocardial injury defined as a rise and/or fall of high-sensitivity cardiac Troponin (hs-cTn) values with at least one value above the 99th percentile Upper Reference Limit at baseline or after presentation.
* Patients scheduled for ICA.
* Written informed consent.

Exclusion Criteria:

* Patients diagnosed with myocardial infarction with ST segment elevation.
* Very High-risk NSTEMI patients according to 2020 ESC Guidelines on Acute Coronary Syndromes:
* Haemodynamic instability
* Cardiogenic shock
* Recurrent/refractory chest pain despite medical treatment
* Life-threatening arrhythmias
* Mechanical complications of MI
* Acute heart failure clearly related to NSTEMI
* ST-segment depression>1mm/6 leads plus ST-segment elevation aVR and/or V1.
* Legally incompetent to provide informed consent
* Participation in another clinical study.
* Regular known contraindications to CMR at time of inclusion such as:
* Severe renal impairment (eGFR < 30 ml / min / 1,73 m2) or on dialysis treatment
* Claustrophobia
* Known pregnancy or breast-feeding patients
* Non MR compatible devices
* Known allergy to Gadolinium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reclassification rate | immediately after invasive coronary angiography
  number of patients in whom the information provided by CMR affects the final diagnosis

SECONDARY OUTCOMES:
Culprit lesion identification | during invasive coronary angiography
  ability of CMR to detect culprit lesion
Revascularization strategy | immediately after invasive coronary angiography
  number of patients in whom CMR affects the revascularization strtegy

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Cardiocentro Ticino, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Data will be avaliable under specific request to Principal Investigator